CLINICAL TRIAL: NCT06900647
Title: Phase I Study to Evaluate the Safety and Preliminary Efficacy of Bortezomib Combined With Cisplatin in Patients With Recurrent or Metastatic Breast Cancer
Brief Title: Bortezomib Plus Cisplatin in Recurrent or Metastatic Breast Cancer
Acronym: BOCIS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Yanxia, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2024-FXY-300
Record Dates: First submitted 2025-03-16; First posted 2025-03-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Breast Cancer; Recurrent Breast Cancer
Keywords: Breast cancer; Bortezomib; Cisplatin
MeSH Terms: conditions — Breast Neoplasms | interventions — Bortezomib; Cisplatin

STUDY DESIGN:
Intervention Model Description: Single-center, non-randomized, open-label, phase I study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dose level 1 (Experimental): In this dose level, all subjects will receive a dose of 1.3m/m2 bortezomib combined with a dose of 50mg/m2 cisplatin.
  Interventions: Drug: Bortezomib (B); Drug: Cisplatin (CDDP)
- Dose level 2 (Experimental): In this dose level, all subjects will receive a dose of 1.5m/m2 bortezomib combined with a dose of 50mg/m2 cisplatin.
  Interventions: Drug: Cisplatin (CDDP); Drug: Bortezomib (B)
- Dose level 3 (Experimental): In this dose level, all subjects will receive a dose of 1.7m/m2 bortezomib combined with a dose of 50mg/m2 cisplatin.
  Interventions: Drug: Cisplatin (CDDP); Drug: Bortezomib (B)
- Dose level 4 (Experimental): In this dose level, all subjects will receive a dose of 1.3m/m2 bortezomib combined with a dose of 75mg/m2 cisplatin.
  Interventions: Drug: Bortezomib (B); Drug: Cisplatin (CDDP)
- Dose level 5 (Experimental): In this dose level, all subjects will receive a dose of 1.5m/m2 bortezomib combined with a dose of 75mg/m2 cisplatin.
  Interventions: Drug: Bortezomib (B); Drug: Cisplatin (CDDP)
- Dose level 6 (Experimental): In this dose level, all subjects will receive a dose of 1.7m/m2 bortezomib combined with a dose of 75mg/m2 cisplatin.
  Interventions: Drug: Bortezomib (B); Drug: Cisplatin (CDDP)

INTERVENTIONS:
Drug: Bortezomib (B) — 1.3mg/m2, IV, D1, D4, D8 and D11, every 3 weeks
  Arms: Dose level 1; Dose level 4
Drug: Cisplatin (CDDP) — 50mg/m2, IV, D1-3, every 3 weeks
  Arms: Dose level 1; Dose level 2; Dose level 3
Drug: Bortezomib (B) — 1.5mg/m2, IV, D1, D4, D8 and D11, every 3 weeks
  Arms: Dose level 2; Dose level 5
Drug: Bortezomib (B) — 1.7mg/m2, IV, D1, D4, D8 and D11, every 3 weeks
  Arms: Dose level 3; Dose level 6
Drug: Cisplatin (CDDP) — 70mg/m2, IV, D1-3, every 3 weeks
  Arms: Dose level 4; Dose level 5; Dose level 6

SUMMARY:
This a phase 1 study to evaluate the safety and preliminary efficacy of cisplatin combined with bortezomib in patients with recurrent or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 years and above with pathologically confirmed recurrent or metastatic advanced breast cancer ;
2. The patient has tumor specimens (formalin-fixed, paraffin-embedded or fresh pre-treated recurrent tumor tissue);
3. Patients who have failed standard treatment in the late stage;
4. At least one measurable lesion;
5. ECOG PS : 0-2 points;
6. Estimated survival period ≥12 weeks;
7. The function level of major organs meets the following standards:

1) The blood routine examination standards must meet: ANC ≥1.5×109/L, PLT ≥75×109/L, Hb ≥85g/L (no blood transfusion and blood products within 14 days, no use of G-CSF and other hematopoietic stimulating factors for correction) 2) Biochemical examinations must meet the following standards: TBIL <1.5×ULN, ALT, AST <2.5×ULN, ALT, AST <5×ULN for patients with liver metastasis, BUN and Cr ≤1×ULN or endogenous creatinine clearance ≥50ml/min (Cockcroft-Gault formula); 8. Women of childbearing age must have taken reliable contraceptive measures, or have undergone a pregnancy test (serum or urine) within 7 days before enrollment, with a negative result, and are willing to use appropriate contraceptive methods during the trial and 8 weeks after the last administration of the trial drug.

9. The subjects voluntarily join this study, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

Any of the following will be considered as meeting the exclusion criteria of the study:

1. Patients with acute active hepatitis B or acute active hepatitis C;
2. Any serious underlying disease, comorbidity and active infection
3. Currently receiving other anti-tumor treatments;
4. History of epilepsy or epileptic-induced condition;
5. Patients who are pregnant or breastfeeding;
6. Those with poor compliance or unable to undergo normal follow-up;
7. Allergic to study drugs;
8. Patients diagnosed with other malignant tumors within 5 years, except for the following: surgically resected non-melanoma skin cancer, adequately treated cervical carcinoma in situ, surgically radically treated ductal carcinoma in situ, or malignant tumors diagnosed 2 years ago with no current evidence of disease and untreated ≤ 2 years before randomization;
9. The researcher determines other situations that may affect the conduct of the clinical study and the determination of the study results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | Within 28 days after the first dose.
  The DLT assessment period is from day 1 to day 21 of the subject's first dose plus 24 hours after the second dose, that is, 22 days.
  Each dose group must first enroll 3 subjects. If no DLT occurs in the first cycle (within 28 days after the first dose), the dose will be increased to the next cohort; if 1 subject develops DLT, 3 subjects will be added to the cohort, and if no DLT occurs in the last 3 subjects, the dose will be increased to the next dose. If 2 or more subjects in 3 or 6 subjects in a dose group develop DLT, the dose escalation will be stopped, and the previous dose of the dose will be the MTD. DLT is defined as a treatment-related adverse event of Grade 3 or higher, based on the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Maximum Tolerated Dose (MTD) | Within 28 days after the first dose.
  If 2 or more subjects in 3 or 6 subjects in a dose group develop DLT, the dose escalation will be stopped , and the previous dose of the dose will be the MTD. If the MTD is not reached in this trial, the researchers will discuss whether to continue the subsequent escalation trial.

SECONDARY OUTCOMES:
Progression- free survival ( PFS ) | Within approximately 48 months.
  PFS assessed by investigators according to RECIST version 1.1 criteria.
Objective Response Rate (ORR) | Within approximately 48 months
  ORR assessed by investigators according to RECIST version 1.1 criteria.
Disease Control Rate (DCR) | Within approximately 48 months
  DCR assessed by investigators according to RECIST version 1.1 criteria.
Area Under the Curve (AUC) | Blood samples for PK analysis were collected within 60 minutes before dosing, at 0.5, 2, 6, 24, 72 hours, and on days 8, 15, and 22 after the start of dosing.
  The area under the plasma concentration-time curve (AUC) will be measured to evaluate the systemic exposure of bortezomib and cisplatin. Blood samples will be collected at specified time points to calculate AUC using non-compartmental analysis.
Maximum Plasma Concentration (Cmax) | Blood samples for PK analysis were collected within 60 minutes before dosing, at 0.5, 2, 6, 24, 72 hours, and on days 8, 15, and 22 after the start of dosing.
  The maximum observed plasma concentration (Cmax) of bortezomib and cisplatin will be determined from the collected blood samples. Cmax reflects the peak concentration of the drug in plasma after administration.
Time to Maximum Plasma Concentration (Tmax) | Blood samples for PK analysis were collected within 60 minutes before dosing, at 0.5, 2, 6, 24, 72 hours, and on days 8, 15, and 22 after the start of dosing.
  The time to reach the maximum plasma concentration (Tmax) will be assessed for bortezomib and cisplatin. Tmax will be determined directly from the plasma concentration-time data.
Half-Life (T1/2) | Blood samples for PK analysis were collected within 60 minutes before dosing, at 0.5, 2, 6, 24, 72 hours, and on days 8, 15, and 22 after the start of dosing.
  The terminal elimination half-life (T1/2) of bortezomib and cisplatin will be calculated using non-compartmental analysis. T1/2 represents the time required for the plasma concentration of the drug to decrease by 50%.

CONTACTS AND LOCATIONS:
Overall Officials: Yan-xia Shi, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical and privacy concerns.

REFERENCES:
- [Background] Shao F, Lyu X, Miao K, Xie L, Wang H, Xiao H, Li J, Chen Q, Ding R, Chen P, Xing F, Zhang X, Luo GH, Zhu W, Cheng G, Lon NW, Martin SE, Wang G, Chen G, Dai Y, Deng CX. Enhanced Protein Damage Clearance Induces Broad Drug Resistance in Multitype of Cancers Revealed by an Evolution Drug-Resistant Model and Genome-Wide siRNA Screening. Adv Sci (Weinh). 2020 Oct 11;7(23):2001914. doi: 10.1002/advs.202001914. eCollection 2020 Dec. PMID 33304752
- [Background] Manasanch EE, Orlowski RZ. Proteasome inhibitors in cancer therapy. Nat Rev Clin Oncol. 2017 Jul;14(7):417-433. doi: 10.1038/nrclinonc.2016.206. Epub 2017 Jan 24. PMID 28117417
- [Background] Irvin WJ Jr, Orlowski RZ, Chiu WK, Carey LA, Collichio FA, Bernard PS, Stijleman IJ, Perou C, Ivanova A, Dees EC. Phase II study of bortezomib and pegylated liposomal doxorubicin in the treatment of metastatic breast cancer. Clin Breast Cancer. 2010 Dec 1;10(6):465-70. doi: 10.3816/CBC.2010.n.061. PMID 21147690
- [Background] Engel RH, Brown JA, Von Roenn JH, O'Regan RM, Bergan R, Badve S, Rademaker A, Gradishar WJ. A phase II study of single agent bortezomib in patients with metastatic breast cancer: a single institution experience. Cancer Invest. 2007 Dec;25(8):733-7. doi: 10.1080/07357900701506573. Epub 2007 Oct 18. PMID 17952740
- [Background] Thaler S, Thiede G, Hengstler JG, Schad A, Schmidt M, Sleeman JP. The proteasome inhibitor Bortezomib (Velcade) as potential inhibitor of estrogen receptor-positive breast cancer. Int J Cancer. 2015 Aug 1;137(3):686-97. doi: 10.1002/ijc.29404. Epub 2015 Jan 8. PMID 25530422
- [Background] Mack PC, Davies AM, Lara PN, Gumerlock PH, Gandara DR. Integration of the proteasome inhibitor PS-341 (Velcade) into the therapeutic approach to lung cancer. Lung Cancer. 2003 Aug;41 Suppl 1:S89-96. doi: 10.1016/s0169-5002(03)00149-1. PMID 12867067
- [Background] Ikezoe T, Yang Y, Saito T, Koeffler HP, Taguchi H. Proteasome inhibitor PS-341 down-regulates prostate-specific antigen (PSA) and induces growth arrest and apoptosis of androgen-dependent human prostate cancer LNCaP cells. Cancer Sci. 2004 Mar;95(3):271-5. doi: 10.1111/j.1349-7006.2004.tb02215.x. PMID 15016328
- [Background] Adams J, Palombella VJ, Sausville EA, Johnson J, Destree A, Lazarus DD, Maas J, Pien CS, Prakash S, Elliott PJ. Proteasome inhibitors: a novel class of potent and effective antitumor agents. Cancer Res. 1999 Jun 1;59(11):2615-22. PMID 10363983
- [Background] Pharoah PD, Day NE, Caldas C. Somatic mutations in the p53 gene and prognosis in breast cancer: a meta-analysis. Br J Cancer. 1999 Aug;80(12):1968-73. doi: 10.1038/sj.bjc.6690628. PMID 10471047
- [Background] Osin PP, Lakhani SR. The pathology of familial breast cancer: Immunohistochemistry and molecular analysis. Breast Cancer Res. 1999;1(1):36-40. doi: 10.1186/bcr11. Epub 1999 Oct 27. PMID 11250681
- [Background] Orlowski RZ, Dees EC. The role of the ubiquitination-proteasome pathway in breast cancer: applying drugs that affect the ubiquitin-proteasome pathway to the therapy of breast cancer. Breast Cancer Res. 2003;5(1):1-7. doi: 10.1186/bcr460. Epub 2002 Aug 14. PMID 12559038
- [Background] Boccadoro M, Morgan G, Cavenagh J. Preclinical evaluation of the proteasome inhibitor bortezomib in cancer therapy. Cancer Cell Int. 2005 Jun 1;5(1):18. doi: 10.1186/1475-2867-5-18. PMID 15929791
- [Background] Lenz HJ. Clinical update: proteasome inhibitors in solid tumors. Cancer Treat Rev. 2003 May;29 Suppl 1:41-8. doi: 10.1016/s0305-7372(03)00082-3. PMID 12738242
- [Background] Cusack JC. Rationale for the treatment of solid tumors with the proteasome inhibitor bortezomib. Cancer Treat Rev. 2003 May;29 Suppl 1:21-31. doi: 10.1016/s0305-7372(03)00079-3. PMID 12738240
- [Background] Adams J. Development of the proteasome inhibitor PS-341. Oncologist. 2002;7(1):9-16. doi: 10.1634/theoncologist.7-1-9. PMID 11854543
- [Background] Kane RC, Farrell AT, Sridhara R, Pazdur R. United States Food and Drug Administration approval summary: bortezomib for the treatment of progressive multiple myeloma after one prior therapy. Clin Cancer Res. 2006 May 15;12(10):2955-60. doi: 10.1158/1078-0432.CCR-06-0170. PMID 16707588
- [Background] Awada A, Albanell J, Canney PA, Dirix LY, Gil T, Cardoso F, Gascon P, Piccart MJ, Baselga J. Bortezomib/docetaxel combination therapy in patients with anthracycline-pretreated advanced/metastatic breast cancer: a phase I/II dose-escalation study. Br J Cancer. 2008 May 6;98(9):1500-7. doi: 10.1038/sj.bjc.6604347. Epub 2008 Apr 29. PMID 18454159

DOCUMENTS (1):
  • Study Protocol (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT06900647/Prot_000.pdf